CLINICAL TRIAL: NCT04543006
Title: Persistence of Neutralizing Antibodies 6 and 12 Months After a Covid-19
Acronym: PANCOLIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: EssaiClinique_PANCOLIN
Record Dates: First submitted 2020-09-08; First posted 2020-09-09 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: neutralizing antibodies; long-term persistence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: sample of patients 6 and 12 months after the acute disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Covid-19 (Other): only arm: Covid-19 proven by PCR
  Interventions: Diagnostic Test: serology

INTERVENTIONS:
Diagnostic Test: serology — blood sample of 10 ml twice (6 and 12 months after the Covid-19)

SUMMARY:
Covid-19 is associated with the onset of anti-SARS-CoV-2 antibodies; in a majority of patients, neutralizing antibodies are detected. However, the long-term persistence of such protective antibodies is not known.

The investigators will explore patients with a proven Covid-19 (positive PCR) 6 and 12 months after the diagnosis to determine whether neutralizing antibodies are still detected.

The investigators will determine whether this persistance varies according to

* the severity of the Covid-19
* a treatment by steroids during the covid-19. This will help to anticipate whether a second wave of infection is possible in a non-naive population.

DETAILED DESCRIPTION:
Covid-19 is associated with the onset of anti-SARS-CoV-2 antibodies; in a majority of patients, neutralizing antibodies are detected. However, the long-term persistence of such protective antibodies is not known.

The investigators will explore adult patients with a proven Covid-19 (positive PCR) 6 and 12 months after the diagnosis to determine whether neutralizing antibodies are still detected.

The investigators will determine whether this persistance varies according to

* the severity of the Covid-19 (3 groups: no oxyegn therapy; oxygen therapy of less than 3L/min; oxygen therapy of 3L/min or more)
* a treatment by steroids during the covid-19. Immunocompromised patients will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* positive SARS-CoV-2

Exclusion Criteria:

* age under 18
* immunocompromised at the onset of Covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-09-08 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
anti-SARS-CoV-2 neutralizing antibody titers | 1 day
  Titer in plamsa of neutralizing anti-SARS-CoV-2 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Epaulard, MD,PhD, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No